CLINICAL TRIAL: NCT01685801
Title: A Pilot Study Testing the Effect of Ivacaftor on Lung Function in Subjects With Cystic Fibrosis, Residual CFTR Function, and FEV1 ≥40% Predicted
Brief Title: Pilot Study Testing the Effect of Ivacaftor on Lung Function in Subjects With Cystic Fibrosis and Residual CFTR Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VX12-770-113
Record Dates: First submitted 2012-09-06; First posted 2012-09-14 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) (Experimental): During the Crossover Period, study drug was administered in 2-week alternating cycles with a minimum of 4-week washout period between Cycle 1 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and Cycle 2 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and between Cycle 2 and the Open-label Period (Day 1 to 57). During the Open-label Period, all participants received ivacaftor.
  Interventions: Drug: Ivacaftor; Drug: Placebo-matched-to-ivacaftor tablet
- Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) (Experimental): During the Crossover Period, study drug was administered in 2-week alternating cycles with a minimum of 4-week washout period between Cycle 1 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and Cycle 2 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and between Cycle 2 and the Open-label Period (Day 1 to 57). During the Open-label Period, all participants received ivacaftor.
  Interventions: Drug: Ivacaftor; Drug: Placebo-matched-to-ivacaftor tablet
- Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) (Experimental): During the Crossover Period, study drug was administered in 2-week alternating cycles with a minimum of 4-week washout period between Cycle 1 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and Cycle 2 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and between Cycle 2 and the Open-label Period (Day 1 to 57). During the Open-label Period, all participants received ivacaftor.
  Interventions: Drug: Ivacaftor; Drug: Placebo-matched-to-ivacaftor tablet
- Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI) (Experimental): During the Crossover Period, study drug was administered in 2-week alternating cycles with a minimum of 4-week washout period between Cycle 1 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and Cycle 2 [(Period 1 - Day 1 to 14) (Period 2 - Day 15 to 29)] and between Cycle 2 and the Open-label Period (Day 1 to 57). During the Open-label Period, all participants received ivacaftor.
  Interventions: Drug: Ivacaftor; Drug: Placebo-matched-to-ivacaftor tablet

INTERVENTIONS:
Drug: Ivacaftor — 150 milligram (mg) tablet orally every 12 hours up to 12 weeks.
  Other Names: Kalydeco, VX-770
Drug: Placebo-matched-to-ivacaftor tablet — Orally every 12 hours up to 4 weeks.

SUMMARY:
This study is a multiple within participant crossover study to evaluate the effect of ivacaftor on lung function in participants aged 12 years and older with cystic fibrosis (CF) who have phenotypic or molecular evidence of residual CF transmembrane conductance regulator (CFTR) function.

DETAILED DESCRIPTION:
CFTR Mutations associated with residual function or defective messenger ribonucleic acid (mRNA) splicing include the following:

R117H, E56K, P67L, D110E, D110H, R117C, R347H, R352Q, A455E, D579G, S945L, L206W, R1070W, F1074L, D1152H, S1235R, D1270N, 2789+5G->A, 3849+10kbC->T, 3272-26A->G, 711+5G->A, 3120G->A, 1811+1.6kbA->G, 711+3A->G, 1898+3A->G, 1898+1G->A, 1717-1G->A, 1717-8G->A, 1342-2A->C, 405+3A->C, 1716G/A 1811+1G->C, 1898+5G->T, 3850-3T->G, IVS14b+5G->A, 1898+1G->T, 4005+2T->C, 621+3A->G, 621+1G->T.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with confirmed diagnosis of CF
* Clinical evidence of residual CFTR function based on any 1 of the following: 1) Clinically documented residual exocrine pancreatic function, 2) Sweat chloride value less than equal to (<=) 80 millimole per liter (mmol/L) at screening, or 3) Age of diagnosis greater than equal to (>=) 12 years and at least 1 copy of a CFTR mutation associated with residual CFTR function or defective mRNA splicing
* FEV1 >= 40 percent (%)
* 12 years of age or older
* Willing to agree to meet the contraception requirements
* Able to swallow tablets

Exclusion Criteria:

* A copy of any of the following CFTR mutations: G551D, G178R, S549N, S549R, G551S, G970R, G1244E, S1251N, S1255P, or G1349D
* Unable to perform spirometry
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before Day 1
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within the 30 days prior to screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nick, MD, Principal Investigator — National Jewish Health
Locations (1):
- Denver, Colorado, United States

REFERENCES:
- [Derived] Nick JA, St Clair C, Jones MC, Lan L, Higgins M; VX12-770-113 Study Team. Ivacaftor in cystic fibrosis with residual function: Lung function results from an N-of-1 study. J Cyst Fibros. 2020 Jan;19(1):91-98. doi: 10.1016/j.jcf.2019.09.013. Epub 2019 Nov 26. PMID 31784217

RESULTS

PARTICIPANT FLOW:
Period: Cycle 1 Period 1 (2 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 6 | 7 | 6
Completed | 5 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Cycle 1 Period 2 (2 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 6 | 7 | 6
Completed | 5 | 6 | 7 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 1 (4 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 6 | 7 | 5
Completed | 5 | 6 | 7 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Cycle 2 Period 1 (2 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 6 | 7 | 5
Completed | 5 | 6 | 7 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Cycle 2 Period 2 (2 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 6 | 7 | 5
Completed | 5 | 5 | 7 | 4
Not Completed | 0 | 1 | 0 | 1
Not completed — Non-compliance with Study Drug | 0 | 1 | 0 | 1
Period: Washout Period 2 (4 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 5 | 7 | 4
Completed | 5 | 5 | 7 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Open-label Period (8 Weeks)
Arm/Group | Ivacaftor, Placebo, Ivacaftor, Placebo (IPIP) | Ivacaftor, Placebo, Placebo, Ivacaftor (IPPI) | Placebo, Ivacaftor, Ivacaftor, Placebo (PIIP) | Placebo, Ivacaftor, Placebo, Ivacaftor (PIPI)
Started | 5 | 5 | 7 | 4
Completed | 5 | 5 | 7 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug (ivacaftor or placebo).
Groups:
- IPIP; IPPI; PIIP; PIPI: Detailed reporting group description is provided in Participant Flow module.
- Total: Total of all reporting groups
Arm/Group | IPIP | IPPI | PIIP | PIPI | Total
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (8.04) | 29.7 (11.66) | 41.4 (13.96) | 33.8 (17.26) | 37.3 (13.86)
Age, Customized [Number; unit: participants]
  less than (<) 20 years | 0 | 1 | 0 | 2 | 3
  20 - 40 years | 1 | 4 | 3 | 2 | 10
  greater than (>) 40 years | 4 | 1 | 4 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 2 | 12
  Male | 2 | 2 | 4 | 4 | 12
Genotype [Number; unit: participants] — All participants were tested for cystic fibrosis transmembrane conductance regulator (CFTR) genotype. Participants with a documented medical history of either a residual function or a messenger ribonucleic acid (mRNA) splice site (Class V) CFTR mutation were reported.
  participants
    mRNA Splice Site (Class V) Mutations | 3 | 3 | 2 | 2 | 10
    Residual Function Mutations | 2 | 3 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Cycle 1 and Cycle 2: Absolute Change From Cycle Baseline In Percent Predicted Forced Expiratory Volume In 1 Second (FEV1) After 2 Weeks of Treatment
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Data was to be reported for each cycle (Cycle 1 and Cycle 2) and as per drug treatment, for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: Cycle 1 baseline, Cycle 1 Day 15 (for Cycle 1 reporting arms); Cycle 2 baseline, Cycle 2 Day 15 (for Cycle 2 reporting arms)
Population: Full analysis set (FAS) population. Here, number of participants analyzed signifies participant evaluable for this outcome measure and "n" signifies participants who were evaluable for the specified category in each arm, respectively.
Measure: Mean (Standard Deviation); unit: Percent predicted of FEV1
Groups:
- Cycle 1: Placebo: Placebo-matched-to-ivacaftor tablet orally every 12 hours for 2 weeks during either in period 1 or 2 of Cycle 1.
- Cycle 1: Ivacaftor: Ivacaftor 150 mg tablet orally every 12 hours for 2 weeks during either in period 1 or 2 of Cycle 1.
- Cycle 2: Placebo: Placebo-matched-to-ivacaftor tablet orally every 12 hours for 2 weeks during either in period 1 or 2 of Cycle 2.
- Cycle 2: Ivacaftor: Ivacaftor 150 mg tablet orally every 12 hours for 2 weeks during either in period 1 or 2 of Cycle 2.
Arm/Group | Cycle 1: Placebo | Cycle 1: Ivacaftor | Cycle 2: Placebo | Cycle 2: Ivacaftor
Number analyzed (Participants) | 24 | 24 | 23 | 23
Percent predicted of FEV1
  Overall (n=24, 24, 23, 23) | 0.5828 (3.67326) | 2.0898 (4.63833) | 0.8495 (4.20641) | 3.6868 (6.13466)
  mRNA Splice Site(ClassV)Mutations (n=10, 10, 9, 9) | -0.5710 (3.39739) | 0.8196 (5.09161) | 1.7132 (3.80933) | 2.0640 (3.55493)
  Residual Function Mutations (n=14, 14, 14, 14) | 1.4069 (3.75842) | 2.9971 (4.24124) | 0.2942 (4.49056) | 4.7300 (7.27436)
Statistical Analysis 1: Comparison: Cycle 1: Placebo vs Cycle 1: Ivacaftor vs Cycle 2: Placebo vs Cycle 2: Ivacaftor; This statistical analysis is for "Overall" category; Test type: Superiority or Other; Posterior Mean = 2.251, 95% CI 2-sided [0.383 to 4.144], Standard Deviation 0.961 — The posterior distribution of overall treatment difference was obtained using the Bayesian hierarchical model and 95% credible interval of the treatment effect (posterior mean) was calculated

2. Secondary Outcome: Cycle 1 and Cycle 2: Absolute Change From Cycle Baseline In Lung Clearance Index (LCI) After 2 Weeks of Treatment
Description: LCI is a measure of ventilation inhomogeneity that is derived from a multiple-breath washout test. The LCI was calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity [FRC]) required to reduce end-tidal concentration of an inert gas to 1/40th of the starting value. Data was to be reported for each cycle (Cycle 1 and Cycle 2) and as per drug treatment. Data was to be reported for each cycle (Cycle 1 and Cycle 2) and as per drug treatment, for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: as for outcome 1
Population: FAS population. Here, number of participants analyzed signifies participant evaluable for this outcome measure and "n" signifies participants who were evaluable for the specified category in each arm, respectively.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cycle 1: Placebo | Cycle 1: Ivacaftor | Cycle 2: Placebo | Cycle 2: Ivacaftor
Number analyzed (Participants) | 23 | 24 | 23 | 22
ratio
  Overall (n=23, 24, 23, 22) | 0.4596 (1.97774) | 0.2822 (3.54741) | 0.4111 (2.39920) | 0.0770 (1.98188)
  mRNA Splice Site(ClassV)Mutations (n=10, 10, 9, 9) | 0.4321 (1.97140) | -0.5306 (1.91374) | 1.0568 (2.12093) | -0.3136 (1.89562)
  Residual Function Mutations (n=13, 14, 14, 13) | 0.4808 (2.06279) | 0.8628 (4.34252) | -0.0039 (2.54929) | 0.3475 (2.06990)

3. Secondary Outcome: Open-label Period: Absolute Change From Open-label Baseline In Percent Predicted Forced Expiratory Volume In 1 Second (FEV1) at Day 57
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Data was to be reported for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: Open-label Baseline, Open-label Day 57
Population: FAS population. Here, number of participants analyzed signifies participant evaluable for this outcome measure and "n" signifies participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: Percent predicted of FEV1
Groups:
- Open-Label Period: Ivacaftor: Ivacaftor 150 mg tablet orally every 12 hours for 8 weeks during the open-label period after washout period 2.
Arm/Group | Open-Label Period: Ivacaftor
Number analyzed (Participants) | 21
Percent predicted of FEV1
  Overall (n=21) | 4.6815 (4.17934)
  mRNA Splice Site(ClassV)Mutations (n=9) | 4.3072 (2.93624)
  Residual Function Mutations (n=12) | 4.9622 (5.02864)

4. Secondary Outcome: Open-label Period: Absolute Change From Open-label Baseline In Lung Clearance Index (LCI) at Day 57
Description: LCI is a measure of ventilation inhomogeneity that is derived from a multiple-breath washout test. The LCI was calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity [FRC]) required to reduce end-tidal concentration of an inert gas to 1/40th of the starting value. Data was to be reported for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: Open-label Baseline, Open-label Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Open-label Period: Ivacaftor: Ivacaftor 150 mg tablet orally every 12 hours in open-label period (8 weeks) after washout period 2.
Arm/Group | Open-label Period: Ivacaftor
Number analyzed (Participants) | 21
ratio
  Overall (n=21) | -1.5687 (2.27137)
  mRNA Splice Site(ClassV)Mutations (n=9) | -1.3459 (2.88447)
  Residual Function Mutations (n=12) | -1.7358 (1.80502)

5. Secondary Outcome: Open-label Period: Absolute Change From Study Baseline In Sweat Chloride at Day 57
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Data was to be reported for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: Study Baseline, Open-label Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Open-label Period: Ivacaftor
Number analyzed (Participants) | 19
millimole per liter (mmol/L)
  Overall (n=19) | -15.74 (14.781)
  mRNA Splice Site(ClassV)Mutations (n=8) | -14.13 (8.254)
  Residual Function Mutations (n=11) | -16.91 (18.493)

6. Secondary Outcome: Open-label Period: Absolute Change From Open-label Baseline In Weight at Day 57
Description: Data was to be reported for overall participants and as per genotype (residual function mutation and mRNA splice site mutation).
Time Frame: Open-label Baseline, Open-label Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Open-label Period: Ivacaftor
Number analyzed (Participants) | 21
kilograms (kg)
  Overall (n=21) | 1.77 (1.906)
  mRNA Splice Site(ClassV)Mutations (n=9) | 2.32 (2.111)
  Residual Function Mutations (n=12) | 1.35 (1.710)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse events (AEs) that started (or increased in severity) from first dose of study drug through completion of Follow-up were considered TEAEs, with exception that if an AE started during a Washout Period and was beyond 14 days from last dose date of preceding cycle, AE was considered as a "Washout Period" AE, and hence not TEAE. A TEAE was attributed to treatment in which it started or to the treatment in second cycling period of previous Crossover Period if it started during a Washout Period. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. Data was to be reported by drug treatment for double-blind crossover period (Cycle 1 up to Washout Period 2) and open-label period.
Time Frame: From first dose of study drug through completion of follow-up visit (up to 26 weeks)
Population: Safety set included all participants who received at least 1 dose of study drug. Here, number of participants analyzed signifies participant evaluable for this outcome measure.
Measure: Number; unit: participants
Groups:
- Crossover Double-blind Period: Placebo: Placebo matched to ivacaftor tablet orally every 12 hours for 2 weeks either during the double blind period 1 or 2 of cycle 1 and cycle 2.
- Crossover Double-blind Period: Ivacaftor: Ivacaftor 150 mg tablet orally every 12 hours for 2 weeks either during the double blind period 1 or 2 of cycle 1 and cycle 2.
Arm/Group | Crossover Double-blind Period: Placebo | Crossover Double-blind Period: Ivacaftor | Open-label Period: Ivacaftor
Number analyzed (Participants) | 24 | 24 | 21
participants
  AEs | 17 | 18 | 20
  SAEs | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through completion of follow-up visit (up to 26 weeks)
Arm/Group | Crossover Double-blind Period: Placebo | Crossover Double-blind Period: Ivacaftor | Open-label Period: Ivacaftor
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24 | 0/21
Other Adverse Events (participants affected / at risk) | 17/24 | 18/24 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Double-blind Period: Placebo (N=24) | Crossover Double-blind Period: Ivacaftor (N=24) | Open-label Period: Ivacaftor (N=21)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover Double-blind Period: Placebo (N=24) | Crossover Double-blind Period: Ivacaftor (N=24) | Open-label Period: Ivacaftor (N=21)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 2
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 | 1 | 2
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Oral viral infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 4
Pyrexia (General disorders) | 1 | 3 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.